CLINICAL TRIAL: NCT00232882
Title: Neurohumoral and Oxidative Influences of Candesartan, Atenolol, Hydrochlorothiazide and Drug Combinations in Essential Hypertensive Patients.
Brief Title: Pharmacodynamic Influences of Candesartan, Atenolol, Hydrochlorothiazide and Drug Combinations in Hypertensive Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Maxime Lamarre-Cliche, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D2452L00003
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Antihypertensive drugs; Clinical Pharmacology; Autonomic nervous system; Renin angiotensin system; Oxidative stress; Inflammatory markers
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Candesartan 16 mg for 4 weeks followed by candesartan 16 mg and hydrochlorothiazide 12.5 mg for 4 weeks
  Interventions: Drug: Candesartan Thiazide
- 2 (Active Comparator): Atenolol 100 mg for 4 weeks followed by atenolol 100 mg + hydrochlorothiazide 12.5 mg for 4 weeks
  Interventions: Drug: Atenolol Thiazide
- 3 (Active Comparator): Thiazide 25 mg for 4 weeks then added with Candesartan 16 mg
  Interventions: Drug: Thiazide Candesartan

INTERVENTIONS:
Drug: Candesartan Thiazide — Candesartan 16 mg for 4 weeks then added hydrochlorothiazide for 4 weeks
  Arms: 1
Drug: Atenolol Thiazide — Atenolol 100 mg for 4 weeks followed by atenolol 100 mg + hydrochlorothiazide 12.5 mg for 4 weeks
  Arms: 2
Drug: Thiazide Candesartan — Thiazide 25 mg for 4 weeks then added with Candesartan 16 mg
  Arms: 3

SUMMARY:
Angiotensin receptor antagonists (ARA), beta-blockers and diuretics do not seem to confer equivalent cardiovascular protection in hard outcomes clinical trials (beta blockers inferior). These results may be explained by differences in their effects on sympathetic activity, oxidative stress, inflammation and renin angiotensin system activation.

How diuretic addition to first line therapy with ARAs and beta-blockers modulates neurohumoral and hemodynamic parameters is not well understood.

The main hypothesis of this study is that an ARA (candesartan) combined or not with a diuretic will not increase sympathetic activity as much as a beta blocker (atenolol). Secondary hypothesis are of similar nature but relate to hemodynamic parameters, oxidative stress markers, inflammatory markers, or the renin angiotensin system.

The main objective of this study is to assess and compare the effects of candesartan and atenolol and their combination with low dose diuretic therapy on the autonomic nervous system, hemodynamic parameters,on oxidative stress, on inflammatory markers, and on the renin-angiotensin system.

Protocol sponsored by Astra Zeneca canada

DETAILED DESCRIPTION:
INTRODUCTION.

Three large clinical trials (STOP-2, HOPE, LIFE) {Hansson, Lindholm, et al. 1999}{Dahlof, Devereux, et al. 2002}{Yusuf, Sleight, et al. 2000} have suggested that drugs that specifically inhibit the renin angiotensin system (RAS) such as ACE inhibitors and Angiotensin Receptor Antagonists (ARA) have blood pressure-independant cardiovascular protecting effects. In the most recent of these studies, the LIFE trial, Losartan-based therapy was superior to atenolol-based therapy in hypertensive patients with left ventricular hypertrophy {Dahlof, Devereux, et al. 2002}. Very recently, the ALLHAT mega-trial suggested that diuretics were as good as ACE inhibitors for cardiovascular protection in hypertensive patients {Major outcomes in moderately hypercholesterolemic, hypertensive patients randomized to pravastatin vs usual care: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT-LLT)}. These apparently conflicting results underline that the mechanisms of cardiovascular protections are not well understood.

ARAs {Balt, Mathy, et al. 2001}{Moreau, Richer, et al. 1993} have sympathoinhibitory properties while beta-blockers induce a small counterregulatory activation of the sympathetic system {Lijnen, Amery, et al. 1979}{Sundlof, Wallin, et al. 1983}{van den Meiracker, Man in 't Veld AJ, et al. 1988}.We have shown recently that telmisartan prevents the increase in NE normally associated with a reduction in BP while there are reports that diuretics tend to stimulate the sympathetic system {Fernandez, Snedden, et al. 1987}{Lake, Ziegler, et al. 1979}. It has been suggested that the superiority of ARAs could be due to their unique effects on the autonomic nervous system.

Angiotensin II receptor antagonism also decrease the oxidative stress induced by angiotensin II and aldosterone {de Cavanagh, Ferder, et al. 1999}{Hornig, Landmesser, et al. 2001}{Onozato, Tojo, et al. 2002}.We have also shown that telmisartan decreases plasma aldosterone and should therefore decrease the oxidative stress associated with a reduction in aldosterone Hydrochlorothiazide and beta-blockers have not been shown to have antioxidative properties {Welch & Wilcox 2001}{Taddei, Virdis, et al. 2001}. It is possible that oxidative stress partly explains the differences between pharmacological agents.

Patients included in high blood pressure clinical trials are randomized to a therapeutic strategy meaning that a stepped care approach is taken. Hypertensive patients frequently need more than one drug for appropriate blood pressure control. Consequently, about half of study patients in these trials end up taking more than one drug during the study. First step therapy is by definition prescribed to all study subjects but second or third step therapy are not as well defined. In the HOPE trial, ramipril was added on top of usual treatment. Most of the patients included in HOPE, LIFE, STOP-2 and ALLHAT took at least one other antihypertensive drug, most frequently a thiazide diuretic. Though results were reported as being ACE inhibitor or ARA based, they mostly reflect a mix of single drug and multiple drugs therapy. Whether the beneficial effects of ARAs and beta-blockers are modulated by thiazide diuretics is presently unknown.

We designed a parallel study that primarily assesses the differences between ARAs, diuretics and beta-blockers. The simultaneously measured parameters reflect renin-angiotensin system activity, sympathetic activity, oxidative stress and systemic inflammation. Secondarily, this study assesses the effects of ARA-diuretic and B-blocker-diuretic combinations on the same parameters.

Results from this study will help to understand the results from the previously mentioned clinical trials. The forced titration from monotherapy to a combination therapy will allow us to measure the influence of drug addition on clinically significant parameters. The simultaneous assessment of renin-angiotensin system activity , sympathetic activity, oxidative stress and systemic inflammation will allow us to observe baseline and pharmacologically-induced associations.

It is also probable that results from this study will have direct clinical influences on high blood pressure therapeutic strategies. Physicians treating hypertension frequently have to choose between increasing drug doses to their maximum or adding a new drug. It is presently unknown if one strategy offers more benefits than the other. This study should provide physicians with clues about the expected benefits for each approach.

GOALS

To assess and compare the effects of candesartan and atenolol combined with low dose diuretic therapy on the autonomic nervous system, on oxidative stress, on inflammatory markers, and on the renin-angiotensin system.

To assess and compare the effects of candesartan and atenolol and low dose diuretic therapy on the autonomic nervous system, on inflammatory markers, on oxidative stress, on inflammatory markers, and on the renin angiotensin system.

PRIMARY OBJECTIVE:

1. To measure and compare the effects candesartan 16 mg + HCT 12.5 mg, candesartan 16 mg + HCT 25.0 mg, and atenolol 100 + 12.5 mg on noradrenalin release 4h post-dose, at trough, and after a 10 minute stand.

SECONDARY OBJECTIVES:

1. To measure and compare the effects candesartan 16 mg + HCT 12.5 mg, candesartan 16 mg + HCT 25.0 mg, and atenolol 100 + 12.5 mg on :

   1. frequency power spectral analysis 4h post-dose, and after a 10 minute stand.
   2. oxidative stress, inflammatory markers and adhesion molecules 4h post-dose.
   3. renin, aldosterone and angiotensin II release/production 4h post-dose and at trough.
   4. Insulin and glucose plasma concentration
2. To measure and compare the influences of HCT 25 mg, candesartan 16 mg, and atenolol 100 mg monotherapy on:

   1. noradrenalin release 4h post-dose, at trough, and after a 10 minute stand.
   2. frequency power spectral analysis 4h post-dose, and after a 10 minute stand.
   3. oxidative stress, inflammatory markers and adhesion molecules 4h post-dose.
   4. renin, aldosterone and angiotensin II release/production 4h post-dose and at trough.
   5. Insulin and glucose plasma concentration

DESIGN

Prospective, randomized, open label, 3 arm, 2 period parallel study preceded by a placebo run in period in non-diabetic patients with essential hypertension.

Titration period: introduction of hydrochlorothiazide (12.5 mg daily), atenolol (50 mg daily), and candesartan (8 mg daily) in the diuretic, beta-blocker and angiotensin receptor blocker groups respectively. First study period (4 weeks), comparison of hydrochlorothiazide 25 mg, atenolol 100 mg, and candesartan 16mg. Second study period (4 weeks), comparison of hydrochlorothiazide 25 mg + candesartan 16 mg, atenolol 100 mg + HCT 12.5 mg, and candesartan 16mg + HCT 12.5 mg. Measurement of study parameters at trough, 4h post-dose and after a 10 minutes stand after placebo and after each study period.

MEASURED STUDY PARAMETERS

1. Blood pressure
2. 24h blood pressure
3. Spectral analysis of heart rate (LF, HF, LF/HF)
4. Plasma

   1. renin
   2. aldosterone
   3. angiotensin II
   4. catecholamines
   5. 8-epi-isoprostane
   6. Thiobarbituric acid reactive substances (TBARS)
   7. nitrotyrosine
   8. interleukin 18
   9. E selectine
   10. C reactive protein
   11. Insulin
   12. glucose
5. Urine

   1. 8-epi-isoprostane
   2. sodium concentration
   3. creatinine concentration

Protocol Sponsored by Astra Zeneca Canada

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate essential hypertension as defined by a morning mean DBP *90 mmHg and * 109 mm Hg, a mean SBP * 200 mm H for two consecutive visits (Visits 2 and 3) during the two-to-four week placebo run-in period,
2. Ability to provide written informed consent.

Exclusion Criteria:

1. Any woman not surgically sterile or menopausal who:

   1. has a positive urine pregnancy test at screening (Visit 1) or baseline (Visit 3)
   2. is breast feeding
2. Pre-menopausal women (last menstruation < 1 year prior to start of run-in period) who:

   1. are not surgically sterile; and/or
   2. are of child-bearing potential and are NOT practicing acceptable means of birth control.
3. Known or suspected secondary hypertension.
4. Known reversible or non-reversible obstructive lung disease (e.g. asthma or COPD).
5. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   1. ALT or AST greater than 2.0 times the upper limit of reference range;
   2. Serum creatinine greater than 150 umol/L.
6. Uncorrected volume depletion.
7. NYHA functional class CHF III-IV (Refer to Appendices).
8. Coronary heart disease needing pharmacological therapy.
9. Stroke within the preceding six months.
10. PTCA within the preceding three months.
11. History of angioedema.
12. Clinically significant sinus bradycardia below 55 beats/min. at randomization.
13. Sustained ventricular tachycardia, atrial fibrillation, or other clinically relevant cardiac arrhythmias as determined by the clinical Investigator.
14. Second or third degree AV block, left bundle branch block or any clinically relevant conduction abnormality as determined by the clinical Investigator.
15. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve.
16. Administration of digoxin.
17. Patients with a fasting glucose > 7.0.
18. Use of antihypertensive agents such as diuretics, ACE inhibitors, angiotensin II antagonists, *- blockers, *-blockers, calcium channel antagonists, direct vasodilators that cannot be stopped for the trial.
19. Administration of other non-antihypertensive medications known to affect blood pressure (e.g., oral corticosteroids, MAO inhibitors, nitrates) at any time during the trial.
20. Chronic use of salt substitutes containing potassium chloride; potassium supplements; extreme dietary restrictions.
21. Uncorrected sodium depletion as defined by a serum sodium level less than 135 mEq/L.
22. Clinically significant hyperkalemia as defined by serum potassium level greater than 5.2 mEq/L. Clinically significant hypokalemia as defined by serum potassium level less than 3.0 mEq/L.
23. Patients receiving any investigational therapy within one month of signing the informed consent form.
24. Known hypersensitivity to any component of candesartan, atenolol or hydrochlorothiazide.
25. Any other clinical condition which, in the opinion of the principal Investigator, would not allow safe completion of the protocol and safe administration of trial medication.
26. Known for allergy to sulfa or heparin
27. Blood donation in the preceding 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Plasma norepinephrine | June 2007

SECONDARY OUTCOMES:
1. Seated blood pressure | June 2007
2. 24h ambulatory blood pressure | June 2007
3. Spectral analysis of heart rate (LF, HF, LF/HF) | June 2007
4. Plasma | December 2007
a. renin | december 2007
b. aldosterone | December 2007
c. angiotensin II | December 2007
d. catecholamines | June 2007
e. 8-epi-isoprostane | December 2007
f. Thiobarbituric acid reactive substances (TBARS) | December 2007
g. nitrotyrosine | December 2007
h. interleukin 18 | December 2007
i. E selectine | December 2007
j. C reactive protein | December 2007
k. Insulin | June 2007
l. glucose | June 2007
5. Urine | June 2007
a. 8-epi-isoprostane | December 2007

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Lamarre-Cliche, MD, Principal Investigator — Institut de Recherches Cliniques de Montreal
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Johnson NP, Kirkeeide RL, Gould KL. Same Lesion, Different Artery, Different FFR!? JACC Cardiovasc Imaging. 2019 Apr;12(4):718-721. doi: 10.1016/j.jcmg.2017.11.029. Epub 2018 Jan 17. No abstract available. PMID 29361484